CLINICAL TRIAL: NCT02876315
Title: The Effect of Combinatorial Nutritional Supplementation on Immune Function in Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Responsible Party: Principal Investigator, Adrian F. Gombart, Associate Professor, Department of Biochemistry and Biophysics, Oregon State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LPI-7531
Record Dates: First submitted 2016-08-11; First posted 2016-08-23 (Estimated); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Vitamin D Deficiency
Keywords: innate immunity; elderly adults; multivitamin supplement; vitamin D; vitamin C; zinc
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Redoxon VI (Experimental): 2 film coated tablets Redoxon VI oral intake daily for 12 weeks
  Interventions: Dietary Supplement: Redoxon VI
- Placebo (Placebo Comparator): 2 film coated tablets placebo oral intake daily for 12 weeks
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Redoxon VI — Each tablet contains:
  Vitamin C (500mg) Vitamin A (1167IU) Vitamin B6 (3.3mg) Vitamin B12 4.8µg) Vitamin D (200IU) Vitamin E (22.5mg) Folic Acid (200µg) Zinc (5mg) Selenium (55µg) Copper (450µg) Iron (2.5mg)
  Other ingredients: Microcrystalline cellulose, magnesium stearate, hydroxypropylmethylcellulose, hydroxypropylcellulose hypromellose, titanium dioxide, microcrystalline cellulose, iron oxide yellow, sodium croscarmellose, and talc
  Other Names: Redoxon Vita Immune
  Arms: Redoxon VI
Dietary Supplement: placebo — Ingredients: Microcrystalline cellulose, magnesium stearate, hydroxypropylmethylcellulose, hydroxypropylcellulose hypromellose, titanium dioxide, microcrystalline cellulose, iron oxide yellow, sodium croscarmellose, and talc
  Arms: Placebo

SUMMARY:
Many older adults do not get enough zinc, vitamin C and vitamin D, and this can be related to decreased ability to fight infection. The purpose of this research study is to determine if taking a multivitamin/mineral supplement every day for 12 weeks will increase the ability of immune cells in blood to kill bacteria.

DETAILED DESCRIPTION:
Vitamins C and D and the mineral zinc are each considered immune modulating micronutrients, but their specific effects on the immune system, especially when used in combination, is relatively unknown. Deficiency in each of these micronutrients is frequently observed in aging adults and may contribute to age-related declines in immune status. Based on prior published studies, the investigators hypothesize that supplementation of older adults with a combination of vitamin C, vitamin D, and zinc will increase the innate ability of neutrophils to kill invading bacteria through a variety of mechanisms, including increased phagocytosis, antimicrobial peptide expression and changes in reactive oxygen species (ROS) production.

Therefore, this study is designed to investigate the effects of Redoxon VI, a supplement consisting of a combination of vitamin C, vitamin D, and zinc on functional markers of the immune system of healthy, older adults when compared to a matched placebo. To accomplish this, the investigators will recruit 40 healthy adults between the ages of 60 and 75 and randomize them to either Redoxon VI or an identical, inactive placebo control supplement to be taken twice a day for 12 weeks.

Since neutrophil-mediated killing is a crucial defense against Staphylococcus aureus infection that declines with age, it will serve as a primary outcome in this study. Using blood collected from individuals before and after supplementation, the investigators will measure the ability of neutrophils to clear S. aureus cells, and compare the killing activity in those individuals receiving the vitamin and mineral supplement to those receiving the placebo. The investigators will confirm these changes in immune cell function by also measuring phagocytic activity in neutrophils, as well as their ability to produce ROS.

As secondary measures of immune function, the investigators will also determine circulating levels of neutrophils, monocytes and lymphocytes, measure cathelicidin antimicrobial peptide (also known as hCAP18/LL-37) levels, and determine changes in circulating levels of inflammatory cytokines.

Based on previous studies, the investigators expect that any increase in functional immune status will correspond to changes in vitamins C, D and zinc status in these individuals. The investigators expect the results from this study to provide the foundation for future studies investigating combinations of supplements on immune function and more extensive studies using these micronutrients to restore declines in immune function observed in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Serum vitamin D level 25-50 nmol/L (10-20 ng/ml), inclusive
* Willing to limit intake of salmon, herring and sardines to one 4-ounce serving per week for 3 weeks prior to and throughout the study.
* Willing to limit intake of oysters, shellfish, liver, beef, lamb and poultry dark meat to one 4-ounce serving per week for 3 weeks prior to and throughout the study.
* Willing to limit intake of citrus fruits and citrus fruit juices to 2 servings per day during the study for 3 weeks prior to and throughout the study.
* Willing to stop taking multivitamins, supplements containing zinc, vitamins C and D, and food/beverage products supplemented with zinc and vitamins C and D for 3 weeks prior to and throughout the study.

Exclusion Criteria:

* Usual dietary intake of zinc >15 mg/day (as determined in Telephone Screening Script)
* Tobacco use, including e-cigarettes, or smoking of any substance (e.g. cannabis) in the past three months or plans to smoke during the study.
* Have undergone a surgical procedure within the past two months or expect a surgical procedure in the next four months.
* Regularly consume more than two alcoholic drinks a day.
* Have participated in another clinical study within the past two months.
* Undergoing UV therapy (e.g. treatment for skin conditions such as psoriasis) or UV tanning.
* Have a significant acute or chronic illness such as cardiovascular disease, kidney or liver disease, diabetes, thyroid or parathyroid disorder, history of cancer less than five years.
* Have had bariatric surgery (e.g. gastric bypass, gastric banding, sleeve gastrectomy, etc.), other gastrointestinal procedure (e.g. cholecystectomy) or disorders (e.g. Crohn's disease, celiac disease, ulcerative colitis)
* Stage II hypertension (either systolic blood pressure > 159 mm Hg or diastolic blood pressure > 99 mm Hg)
* BMI < 18.5 or > 29.9
* Diagnosis of hypervitaminosis A, hypervitaminosis D, or hypercalcemia
* Have received an organ or tissue transplant
* Have eczema, atopic dermatitis, or psoriasis
* Have or have had allergy to medications or foods, seasonal allergies or allergic asthma after age 18 (childhood asthma/allergies not exclusionary)
* Diagnosis of an autoimmune disorder (e.g. lupus, rheumatoid arthritis, multiple sclerosis, etc.) or HIV positive status.
* Currently taking or using any of the following medications:

  * Topical medications containing retinoids
  * Desferioxamine
  * Disulfiram
  * Warfarin
  * Vitamin D analogs
  * Vitamin A analogs
  * Cholestyramine
  * Orlistat
  * Mineral oil (oral intake)
  * Thiazide diuretics
  * Calcium channel blockers
  * Phenobarbital or phenytoin or other anticonvulsants
  * Estrogen replacement therapy
  * Leukotriene receptor antagonists
  * Immunosuppressant/anti-rejection drugs
  * Oral corticosteroids

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
S. aureus clearance from whole blood | 12 weeks
  Determine the clearance of S. aureus by whole blood from individuals before and after treatment with Redoxon VI or placebo using a whole blood killing functional assay

SECONDARY OUTCOMES:
Determine phagocytic activity of neutrophils by measuring uptake of fluorescently labeled Escherichia coli using flow cytometry | 12 weeks
  Determine phagocytic activity of neutrophils before and after treatment. The investigators will measure phagocytic activity by quantifying the uptake of pHrodoTM Red-labeled Escherichia coli (LifeTechnologies, Carlsbad, CA) by fluorescence activated cell sorting (FACS). The amount of bacteria taken-up by the neutrophils will be determined by mean fluorescence of all cells.
Total ROS generation by neutrophils | 12 weeks
  Determine total ROS generation by neutrophils before and after treatment.
Number of neutrophils, monocytes and lymphocytes | 12 weeks
  Determine the number of circulating neutrophils, monocytes and lymphocytes in blood of individuals before and after treatment.
hCAP18 levels in neutrophils, monocytes and serum | 12 weeks
  Determine hCAP18 levels in neutrophils, monocytes and sera from individuals before and after treatment.
Serum levels of inflammatory cytokines | 12 weeks
  Determine levels of inflammatory cytokines in sera from individuals before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian F Gombart, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fantacone ML, Lowry MB, Uesugi SL, Michels AJ, Choi J, Leonard SW, Gombart SK, Gombart JS, Bobe G, Gombart AF. The Effect of a Multivitamin and Mineral Supplement on Immune Function in Healthy Older Adults: A Double-Blind, Randomized, Controlled Trial. Nutrients. 2020 Aug 14;12(8):2447. doi: 10.3390/nu12082447. PMID 32823974